CLINICAL TRIAL: NCT02942316
Title: Pupillary Dilation Reflex (PDR) Evaluation During General Anesthesia: a Pilot Study
Brief Title: Pupillary Dilation Reflex (PDR) Evaluation During General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/40/410
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Heart Rate; Reflex, Pupillary; Monitoring, Intraoperative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pupil dilation reflex measurement (Experimental): Four measurements of PDR during surgery at standardized times
  Interventions: Device: Pupil dilation reflex measurement

INTERVENTIONS:
Device: Pupil dilation reflex measurement — Pupillometry (PDR) at four standardized times perioperatively
  * after induction, before opioid administration
  * after opioid administration, steady state
  * surgical incision
  * end of procedure

SUMMARY:
In this study, the pupillary dilation reflex is measured as a nociceptive indicator during elective abdominal surgery under general anesthesia.

DETAILED DESCRIPTION:
An infrared camera of the video pupillometer measures the pupillary dilation reflex (PDR) in response of a nociceptive stimulus. This autonomic reflex, parasympathetic mediated in sedated patients, can be generated by various pain stimuli (built in standardized protocol, surgical incision, …) The PDR is a robust reflex, even in patients under general anesthesia, and provides a potential evaluation of the autonomous circuit within the nociceptive evaluation based on pupil dilation upon A-delta and C fibers in both electrical or mechanic stimulation. This mono-centric project involving American Society of Anesthesiologists (ASA) classification I-II patients undergoing elective abdominal surgery under general anesthesia are recruited. Enrolled patients perioperative undergo PDR measurements at four different standardized times.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled abdominal surgery
* ASA I-II

Exclusion Criteria:

* History of eye deformity, invasive ophthalmologic surgery, impaired pupil reflex in advance
* Kown cranial nerve(s) deficit
* Infection of the eye
* Predicted difficult airway management (DAF Guidelines)
* Chronic opioid use (>3 months)
* Ongoing treatment with beta-blockers, dopamine antagonists, topical atropine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pupillary Reflex Dilation | Perioperative phase
  Pupillary Reflex Dilation is measured four times intraoperatively as a possible indicator of success of analgesia

SECONDARY OUTCOMES:
Patient Movement | Perioperative phase
  Patient movement during surgery as a common used indicator for pain
Vital signs | Perioperative phase
  Increased vital signs (heart rate, blood pressure) during surgery as a common used indicator for pain

CONTACTS AND LOCATIONS:
Overall Officials: Robert Slappendel, MD, PhD, Study Director — University Hospital, Antwerp; Michiel Baeten, MD, Principal Investigator — University Hospital, Antwerp; Davina Wildemeersch, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5931178/